CLINICAL TRIAL: NCT03989271
Title: Impact of Quercetin on Inflammatory and Oxidative Stress Markers in COPD
Brief Title: Biological Effects of Quercetin in COPD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Quercegen Pharmaceuticals (Industry); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Umadevi Sajjan, Associate Professor, Temple University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25738; R33AT009991 (NIH)
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Inflammation; Oxidative stress; Plant polyphenol; Flavonols
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation | interventions — Quercetin

STUDY DESIGN:
Intervention Model Description: Double blinded placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization codes will be generated by a study statistician at the begnining of the study and is provided to research pharmacist who will be dispensing the study drugs. The study drug bottles will be numbered with no information about the study drug. The randomization codes will not be revealed until all the data is collected and analyzed. Both placebo and quercetin will be similarly packaged and will have similar color, taste and texture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Quercetin (Active Comparator): Quercetin 2000 mg/day Quercetin is provided as orange flavored soft chews and each chew will have 250 mg of quercetin Quercetin will be administered orally twice daily, one half dose (4 chews) in the morning after breakfast and one half dose (4 chews) in the evening after dinner for six months.
  Interventions: Drug: Quercetin
- Placebo (Placebo Comparator): Placebo is also provided as soft chews that is similar to quercetin in color, taste and texture and will contain all the stabilizers and the inactive ingredients that is present in the quercetin chews.
  Placebo will be administered orally twice daily, one half dose (4 chews) in the morning after breakfast and one half dose (4 chews) in the evening after dinner for six months.
  Interventions: Drug: Quercetin

INTERVENTIONS:
Drug: Quercetin — Placebo
  Other Names: placebo

SUMMARY:
This study determines whether quercetin supplementation reduces the inflammation and oxidative stress markers in patients with chronic obstructive pulmonary disease. It is small study with 8 subjects receive quercetin 2000 mg/day and 4 subjects receive placebo.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a progressive lung disorder and affects millions of people globally. Although the exact mechanisms of pathogenesis of this disease are not well-understood, the general consensus is that oxidative stress and inflammation induced by exposure to cigarette smoke or other environmental or occupational hazards are responsible for development of COPD. Therefore, therapies aimed at decreasing oxidative stress and inflammation constitutes an important component of treating COPD.

The current pharmacological therapies may provide temporary symptom relief, reduce acute exacerbations and hospitalizations, but are associated with side effects. Therefore complementary method of treatment with potentially fewer side effects and relatively well-tolerated provide promising alternative. One such compound is quercetin, which is plant polyphenol and is present in variety of foods that we consume. Quercetin has potent antioxidant and anti-inflammatory properties and reduces oxidative stress and inflammation in a preclinical model of COPD. Quercetin exerts it antioxidant properties not only by neutralizing free radical species, but also by enhancing the expression of antioxidant enzymes. Similarly, quercetin inhibits various protein and lipid kinases by competing for adenosine triphosphate (ATP) binding sites thus reducing the inflammatory pathways.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with COPD, 40 - 80 yrs of age
* Post-bronchodilator forced expiratory volume (FEV)1/forced vital capacity (FVC) ratio 0.7, FEV1% predicted between 40 to 70
* Both active and ex-smokers with at least 10 pack-years history of smoking
* COPD patients taking H2 antagonists, loperamide or loratadine and willing to stop during the study period

Exclusion Criteria:

* Known allergy/sensitivity to quercetin
* Subjects with primary current diagnosis of asthma
* Upper respiratory tract infection within two weeks of the screening visit
* Acute bacterial infection requiring antibiotics within two weeks of screening
* Emergency treatment or hospitalization within one month of screening for any reasons
* Unwillingness to stop flavonoid supplementation
* Dietary intake exceeding or averaging 150 mg quercetin daily as assessed by Bioflavonoid Food and Supplement Screener
* Daily warfarin or cyclosporine (Neoral, Sandimmune)
* Subjects taking H2 antagonists (cimetidine, ranitidine), loperamide (Imodium) or loratadine and not willing to stop during study period
* Lung cancer history or undergoing chemo- or radiation therapy
* Inflammatory bowel disease
* Subjects with no detectable levels of inflammatory CRP or SP-D in blood and/or IL-

  1β or 8-isoprostane in the exhaled breath condensate
* Women of child-bearing age and unwilling to take pregnancy test
* Child-bearing age, who are unwilling to use adequate contraception or abstain during the course of the study.
* Pregnant or lactating mothers

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress markers | six months
  8-isoprostane
Inflammatory markers | six months
  Interleukin (IL)-1beta, IL-8, in bronchoalveolar lavage and C-reactive protein (CRP) and surfactant protein (SP)-D in serum

SECONDARY OUTCOMES:
Quercetin | six months
  Levels of quercetin in blood and lung

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Marchetti, D.O., Principal Investigator — Temple University
Locations (1):
- Nathaniel Marchetti, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ganesan S, Faris AN, Comstock AT, Chattoraj SS, Chattoraj A, Burgess JR, Curtis JL, Martinez FJ, Zick S, Hershenson MB, Sajjan US. Quercetin prevents progression of disease in elastase/LPS-exposed mice by negatively regulating MMP expression. Respir Res. 2010 Sep 28;11(1):131. doi: 10.1186/1465-9921-11-131. PMID 20920189
- [Result] Farazuddin M, Mishra R, Jing Y, Srivastava V, Comstock AT, Sajjan US. Quercetin prevents rhinovirus-induced progression of lung disease in mice with COPD phenotype. PLoS One. 2018 Jul 5;13(7):e0199612. doi: 10.1371/journal.pone.0199612. eCollection 2018. PMID 29975735
- [Result] Ganesan S, Faris AN, Comstock AT, Wang Q, Nanua S, Hershenson MB, Sajjan US. Quercetin inhibits rhinovirus replication in vitro and in vivo. Antiviral Res. 2012 Jun;94(3):258-71. doi: 10.1016/j.antiviral.2012.03.005. Epub 2012 Mar 23. PMID 22465313
- [Derived] McCluskey ES, Liu N, Pandey A, Marchetti N, Kelsen SG, Sajjan US. Quercetin improves epithelial regeneration from airway basal cells of COPD patients. Respir Res. 2024 Mar 11;25(1):120. doi: 10.1186/s12931-024-02742-0. PMID 38468259
- [Derived] McCluskey ES, Liu N, Pandey A, Marchetti N, Sajjan U. Quercetin improves epithelial regeneration from airway basal cells of COPD patients. Res Sq [Preprint]. 2023 Jul 25:rs.3.rs-3185241. doi: 10.21203/rs.3.rs-3185241/v1. PMID 37546740
- See also: Phase I clinical trials to determine the safety of quercetin supplementation in COPD — http://clinicaltrials.gov/ct2/show/NCT01708278